CLINICAL TRIAL: NCT03958500
Title: Problem of Safety of Anastomosis in Colorectal Surgery and Search for the Solutions
Brief Title: The Problem of Colorectal Anastomosis Safety
Acronym: ANSCRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Collaborators: Vilnius University hospital Santaros klinikos, Vilnius, Lithuania (Unknown); National Cancer Center Affiliate of Vilnius University Hospital Santaros Klinikos (Other)
Responsible Party: Principal Investigator, Marius Kryzauskas, Principal investigator, Vilnius University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019/3-1116-608
Record Dates: First submitted 2019-04-17; First posted 2019-05-22 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Cancer; Colorectal Carcinoma; Colorectal Neoplasms; Colorectal Adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comprehensive anastomotic testing (Experimental): All patients undergo:
  1. Indocyanine green fluorescent angiography intraluminally and intraperitoneally
  2. Air leak test
  3. Methylene blue test
  Interventions: Procedure: Indocyanine green fluorescent angiography intraluminally and intraperitoneally

INTERVENTIONS:
Procedure: Indocyanine green fluorescent angiography intraluminally and intraperitoneally — The use of indocyanine green fluorescent angiography to check bowel and anastomosis viability in standard low anterior rectal anastomosis
  Other Names: Air leak test; Methylene blue test

SUMMARY:
This is a prospective cohort pilot study. The investigators are planning to develop an original, standardized colorectal anastomosis inspection method, which will systemically inspect the anastomosis vascularity using the indocyanine green fluorescent angiography intraluminally and intraperitoneally, the air leak test, the methylene blue test, the tension in the anastomosis inspection, patients' risk factors scale sum. The summarized evaluation will determine the final anastomotic leak risk.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 year
* signed written consent
* a colorectal anastomosis lower 15 cm from anal verge
* elective surgery

Exclusion Criteria:

* allergy to indocyanine green dye
* pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Rate of anastomotic leakage | 0 to 60 days
  The number of patients, who had clinical or radiological anastomotic leakage. Proctography will be performed 6-8 days and 4-6 weeks after the primary operation.

SECONDARY OUTCOMES:
Quality of life before and after the operation | 0 to 60 days
  Using low anterior resection syndrome score (the LARS score - simple 5 question questionnaire). LARS score is a tool consisting of five items, which are as follows: incontinence due to flatus (score range from 0 to 7), incontinence due to liquid stools (score range from 0 to 3), frequency of bowel movements (score range from 0 to 5), clustering (score range from 0 to 11) and urgency (score range from 0 to 16). The severity of each item is calculated on a scale ranging from 0 to 42, with a score of 0-20 (no LARS), 21-29 (minor LARS) and 30-42 (major LARS).
Quality of life before and after the operation | 0 to 60 days
  Using QLQ-C30 questionnaire. To compare change in Quality of Life, as defined by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30 (Version 3)) before operation and 4-6 weeks after the operation.
  The EORTC QLQ-C30 (Version 3) uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.
  The EORTC QLQ-C30 (Version 3) uses for the questions 29 and 30 a 7-points scale. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. First of all, raw score has to be calculated with mean values. Afterwards linear transformation is performed to be comparable. More points are considered to have a better outcome.
Reoperation rate | 0 to 60 days
  Patients, who needed re-interventions
Intraoperative test leakage | 0 to 600 minutes
  Leakage rate detected intraoperatively after anastomosis testing
Time of anastomosis testing | 0 to 600 minutes
  Time from the start of the anastomosis testing till the end
Operation time | 0 to 600 minutes
  Time from the start of the operation until the end of the operation
90 days mortality | 0 to 90 days
  the mortality of the patients after the operation
Timing of anastomosis leakage | 0 to 60 days
  In days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Eligijus Poskus, prof., Principal Investigator — Vilnius University, Vilnius, Lithuania
Locations (2):
- Lithuania (2):
  - National Cancer Institute, Vilnius, Lithuania, Vilnius
  - Vilnius University hospital Santaros klinikos, Vilnius

REFERENCES:
- [Derived] Kryzauskas M, Poskus E, Dulskas A, Bausys A, Jakubauskas M, Imbrasaite U, Makunaite G, Kuliavas J, Bausys R, Stratilatovas E, Strupas K, Poskus T. The problem of colorectal anastomosis safety. Medicine (Baltimore). 2020 Jan;99(2):e18560. doi: 10.1097/MD.0000000000018560. PMID 31914032
- See also: Protocol — https://journals.lww.com/md-journal/Fulltext/2020/01100/The_problem_of_colorectal_anastomosis_safety.23.aspx
- See also: Study results — https://link.springer.com/article/10.1007/s00464-022-09093-1